CLINICAL TRIAL: NCT00394329
Title: Childhood Asthma Research and Education (CARE) Network Trial - Treating Children to Prevent Exacerbations of Asthma (TREXA)
Brief Title: (CARE Network Trial - Treating Children to Prevent Exacerbations of Asthma (TREXA)
Acronym: TREXA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 445; 5U10HL064313 (NIH); 5U10HL064288 (NIH); 5U10HL064305 (NIH); 5U10HL064295 (NIH); 5U10HL064287 (NIH); 5U10HL064307 (NIH)
Record Dates: First submitted 2006-10-30; First posted 2006-11-01 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol; Procaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Daily ICS + Rescue ICS (Experimental): Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) one puff bid + beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed + albuterol sulfate HFA (ProAir®™ 90 mcg Inhalation Aerosol) rescue puffs as needed
  Interventions: Drug: Beclomethasone dipropionate; Drug: Albuterol sulfate
- Daily ICS (Active Comparator): Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) one puff bid + albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Interventions: Drug: Beclomethasone dipropionate; Drug: Albuterol sulfate
- Rescue ICS (Experimental): Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed + albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Interventions: Drug: Beclomethasone dipropionate; Drug: Albuterol sulfate
- Placebo (Placebo Comparator): Albuterol sulfate administered via a hydrofluoroalkane (HFA) inhaler (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Interventions: Drug: Albuterol sulfate

INTERVENTIONS:
Drug: Beclomethasone dipropionate — Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) one puff bid
  Other Names: QVAR®
  Arms: Daily ICS; Daily ICS + Rescue ICS
Drug: Beclomethasone dipropionate — Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed
  Other Names: QVAR®
  Arms: Daily ICS + Rescue ICS; Rescue ICS
Drug: Albuterol sulfate — Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Other Names: ProAir®

SUMMARY:
Asthma is a common, serious illness among children in the United States. It can be effectively controlled through the use of preventative medications and "rescue" medications, which are used to control symptoms. This study will evaluate the impact and severity of asthma exacerbations that occur in children with mild persistent asthma who are receiving various combinations of medications for daily and rescue use.

DETAILED DESCRIPTION:
Almost 9 million children in the United States have asthma, and it is a leading cause of hospitalizations and school absenteeism. Common asthma symptoms include wheezing, shortness of breath, chest tightness, and coughing. While there is no cure for asthma, most children who receive proper treatment are able to control symptoms and lead a normal life. Asthma is commonly treated with two types of medications: long-term control medication, such as inhaled corticosteroids (ICS), which is taken on a regular schedule to prevent symptoms and keep asthma under control, and quick-relief, or "rescue" medication, such as albuterol, which is used on an as-needed-basis with the onset of symptoms or an asthma attack. The purpose of this study is to assess the impact and severity of asthma exacerbations that occur in children with mild persistent asthma who are receiving ICS on a daily basis plus ICS and albuterol as rescue medications.

This study will begin with a 4-week screening period during which participants will be monitored while they use an inhaler with a low dose of ICS medication. Study visits will occur at study entry and Week 4. Participants will undergo a physical examination, lung function and airway pressure testing, and blood collection. At the Week 4 study visit, participants will be randomly assigned to one of the following four groups for 44 weeks of treatment:

* Group 1 will take ICS twice a day and ICS plus albuterol as rescue medication
* Group 2 will take ICS twice a day and placebo ICS plus albuterol as rescue medication
* Group 3 will take placebo ICS twice a day and ICS plus albuterol as rescue medication
* Group 4 will take placebo ICS twice a day and placebo ICS plus albuterol as rescue medication

Each participant will receive three inhalers with their assigned medication. One inhaler will be used twice daily throughout the study. The other two inhalers will be used consecutively on an as-needed-basis as rescue medication. Study visits will occur at Weeks 8, 16, 24, 32, 40, and 48. A physical examination, blood collection, and lung function and airway pressure testing will occur at selected visits. Questionnaires to assess quality of life and asthma control will also be completed. A methacholine challenge test will be completed at some study visits. This test artificially triggers an asthma attack to determine the severity of an individual's asthma. Throughout the study, participants will record asthma symptoms and rescue medication usage in a daily diary.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform reproducible spirometry according to American Thoracic Society (ATS) criteria
* History of asthma symptoms that are adequately controlled in the 4 weeks prior to study entry, and meets at least one of the following criteria:

  1. History of mild persistent asthma symptoms (on average greater than 2 days per week with symptoms or albuterol use for symptoms or greater than 2 night-time awakenings per month during the year prior to study entry) and has been treated with a single-controller inhaled corticosteroid (ICS) dose less than or equal to 160 mcg per day of a beclomethasone-equivalent or a leukotriene receptor antagonist (LTRA) (in an age-appropriate dose) for the 4 weeks prior to study entry; individuals treated with a combination controller therapy (e.g. ICS+LTRA or ICS+long-acting beta-agonist (LABA)) in the past 8 weeks will not be eligible
  2. Not currently being treated with ICS, a history of mild persistent asthma, and 1 to 2 exacerbations in the year prior to study entry (but none in the 3 months prior to study entry)
* Forced expiratory volume in one second (FEV1) reversibility of greater than or equal to 12% following bronchodilator administration (4 puffs); individuals who do not meet this requirement may qualify for enrollment if their methacholine provocative concentration at 20% (PC20) is less than or equal to 12.5 milligrams per milliliter (mg/ml)
* History of clinical varicella or varicella vaccine; individuals needing the vaccine may receive it from their primary care physician prior to study entry
* Ability of parent to provide informed consent; verbal assent must be obtained from children less than 7 years of age and written assent must be obtained from children between 7 and 18 years of age
* If female, willing to use an effective form of contraception

Participants will be eligible for the 44 weeks of treatment if, after the 4-week screening period, their asthma remains controlled, and they demonstrate at least 80% predicted pre-bronchodilator FEV1. Participants must meet ALL of the criteria stated below during the 8-week screening period to continue in the study:

* Meets the definition of acceptable asthma control, which is NOT having one or more of the following during ANY 2-week period:

  1. On average, on more than 2 days per week, experiences one or more of the following:

     1. Diary-reported symptoms
     2. The use of inhaled bronchodilator (not including pre-exercise)
     3. Peak flows in the yellow zone (less than 80% of personal best defined as based on peak expiratory flow (PEF) value obtained at study visit 1
  2. More than 1 night-time awakening due to asthma
* Demonstrates adherence with taking study medications (at least 75% of scheduled doses), rescue medications (using both rescue inhalers for at least 75% of rescue doses), and completing patient diaries (at least 75% of days)
* Pre-bronchodilator FEV1 greater than or equal to 80% predicted at study visits 2 and 3
* Agrees to not use a spacer with beclomethasone/placebo study and rescue medications

NOTE: In January 2008, the Data and Safety Monitoring Board (DSMB) approved changes in the TREXA eligibility criteria, by which neither FEV1 reversibility ≥ 12% nor a participant's methacholine PC20 ≤ 12.5 mg/ml were required for randomization.

Exclusion Criteria:

* Corticosteroid treatment for any condition prior to study entry within the following defined timepoints:

  1. Oral - Use within 2-week period of the screening visit
  2. Injectable - Use within 2-week period of the screening visit
  3. Nasal corticosteroids may be used at any time during the study at the discretion of the study investigator or primary care physician
* Current or prior use of medications known to significantly interact with corticosteroid disposition (within a 2-week period of study visit 1), including but not limited to carbamazepine, erythromycin or other macrolide antibiotics, phenobarbital, phenytoin, rifampin, or ketoconazole
* Pre-bronchodilator FEV1 less than 60% predicted at study visit 1
* Any hospitalization for asthma in the year prior to study entry
* Presence of chronic or active lung disease other than asthma
* Significant medical illness other than asthma, including thyroid disease, diabetes mellitus, Cushing's disease, Addison's disease, hepatic disease, or concurrent medical problems that could require oral corticosteroids during the study
* History of cataracts, glaucoma, or any other medical disorder associated with an adverse effect to corticosteroids
* Any asthma exacerbation in the past 3 months or more than 2 in the past year.
* History of a life-threatening asthma exacerbation requiring intubation, mechanical ventilation, or resulting in a hypoxic seizure
* History of adverse reactions to ICS preparations or any of its ingredients
* Receiving hyposensitization therapy other than an established maintenance regimen (continuous regimen for at least 3 months)
* Pregnant or breastfeeding
* Cigarette smoking or smokeless tobacco use in the year prior to study entry
* Refusal to consent to a genotype evaluation
* Current participation or participation within 1 month of study entry in another investigational drug trial
* Evidence that the family may be unreliable or nonadherent, or may move from the clinical center area before study completion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Actual)
Dates: Start 2006-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Mauger, PhD, Principal Investigator — Penn State College of Medicine; Stanley J. Szefler, MD, PhD, Principal Investigator — National Jewish Health; Robert F. Lemanske, Jr., MD, Principal Investigator — University of Wisconsin, Madison; Robert S. Zeiger, MD, PhD, Principal Investigator — Kaiser Permanente Medical Center; Robert C. Strunk, MD, Principal Investigator — Washington University School of Medicine; Fernando D. Martinez, MD, Principal Investigator — University of Arizona College of Medicine; Lynn M. Taussig, MD, Study Chair — University of Denver
Locations (6):
- United States (6):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Los Angeles, Kaiser Permanente Allergy Department, Los Angeles, California
  - Kaiser Permanente Medical Center, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Result] Martinez FD, Chinchilli VM, Morgan WJ, Boehmer SJ, Lemanske RF Jr, Mauger DT, Strunk RC, Szefler SJ, Zeiger RS, Bacharier LB, Bade E, Covar RA, Friedman NJ, Guilbert TW, Heidarian-Raissy H, Kelly HW, Malka-Rais J, Mellon MH, Sorkness CA, Taussig L. Use of beclomethasone dipropionate as rescue treatment for children with mild persistent asthma (TREXA): a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Feb 19;377(9766):650-7. doi: 10.1016/S0140-6736(10)62145-9. Epub 2011 Feb 14. PMID 21324520
- [Derived] Kew KM, Flemyng E, Quon BS, Leung C. Increased versus stable doses of inhaled corticosteroids for exacerbations of chronic asthma in adults and children. Cochrane Database Syst Rev. 2022 Sep 26;9(9):CD007524. doi: 10.1002/14651858.CD007524.pub5. PMID 36161875
- See also: Click here for the Childhood Asthma Research and Education (CARE) Network web site — http://www.asthma-carenet.org

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Daily ICS + Rescue ICS: Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) one puff bid + beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed + albuterol sulfate HFA (ProAir®™ 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate: Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) one puff bid
  Albuterol sulfate : Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate : Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed
- B: Daily ICS: Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) one puff bid + albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate: Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) one puff bid
  Albuterol sulfate : Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
- C: Rescue ICS: Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed + albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Albuterol sulfate: Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate: Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed
- D: Placebo: Albuterol sulfate administered via a hydrofluoroalkane (HFA) inhaler (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Albuterol sulfate: Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
Period: Overall Study
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Started | 71 | 72 | 71 | 74
Completed | 63 | 63 | 58 | 50
Not Completed | 8 | 9 | 13 | 24

BASELINE CHARACTERISTICS:
Groups:
- A: Daily ICS + Rescue ICS: Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) one puff bid + beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed + albuterol sulfate HFA (ProAir®™ 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate: Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) one puff bid
  Albuterol sulfate: Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate: Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) rescue puffs as needed
- B: Daily ICS: Beclomethasone dipropionate administered via a hydrofluoroalkane (HFA) inhaler (QVAR® 40 mcg Inhalation Aerosol) one puff bid + albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
  Beclomethasone dipropionate: Beclomethasone dipropionate HFA (QVAR® 40 mcg Inhalation Aerosol) one puff bid
  Albuterol sulfate: Albuterol sulfate HFA (ProAir® 90 mcg Inhalation Aerosol) rescue puffs as needed
- Total: Total of all reporting groups
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo | Total
Number analyzed (Participants) | 71 | 72 | 71 | 74 | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 71 | 72 | 71 | 74 | 288
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (3.1) | 10.8 (3.5) | 10.4 (2.8) | 10.4 (3.2) | 10.7 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 34 | 33 | 129
  Male | 39 | 42 | 37 | 41 | 159
Region of Enrollment [Number; unit: participants]
  United States | 71 | 72 | 71 | 74 | 288

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing an Asthma Exacerbation That Requires Systemic Corticosteroid Therapy
Time Frame: Measured during the 44-week treatment period
Population: All randomized participants were included in the time-to-event analysis
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
participants | 22 [15 to 31] | 20 [13 to 29] | 25 [17 to 33] | 36 [27 to 45]
Statistical Analysis 1: Comparison: A: Daily ICS + Rescue ICS vs D: Placebo; Test type: Superiority or Other; p = 0.066, Regression, Cox — Hochberg adjustment was applied to the p-value to account for each of three active group comparisons to the placebo group. The unadjusted p-value is 0.033; Cox Proportional Hazard = 0.56, 95% CI 2-sided [0.32 to 0.96], Standard Error of Mean 0.28

2. Secondary Outcome: Change Between Week 44 and Week 0 in the Asthma Control Days
Time Frame: An asthma control day was determined daily during each of the 44-week treatment periods. The primary analysis constructed the change between week 14 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: proportion of asthma control days
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
proportion of asthma control days | -0.006 (0.03) | -0.021 (0.03) | -0.064 (0.03) | -0.034 (0.03)

3. Secondary Outcome: Change Between Week 44 and Week 0 in Rescue Albuterol Puffs Per Day
Time Frame: Rescue albuterol puffs were measured daily during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: count of the number of puffs per day
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
count of the number of puffs per day | 0.26 (0.11) | 0.24 (0.08) | 0.26 (0.09) | 0.18 (0.09)

4. Secondary Outcome: Change Between Week 44 and Week 0 in the Pre-bronchodilator Forced Expiratory Volume in One Second (FEV!)
Time Frame: Pre-bronchodilator FEV1 was measured on seven occasions during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
liters | 0.104 (0.04) | 0.113 (0.04) | 0.097 (0.05) | 0.063 (0.04)

5. Secondary Outcome: Change Between Week 44 and Week 0 in the Morning Peak Expiratory Flow Rate (PEFR)
Time Frame: Morning PEFR was measured daily during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: liters per minute
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
liters per minute | 17.7 (4.4) | 16.3 (4.8) | 16.5 (4.9) | 21.1 (5.4)

6. Secondary Outcome: Change Between Week 44 and Week 0 in the Evening Peak Expiratory Flow Rate Variability (PEFR)
Time Frame: Evening PEFR was measured daily during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: liters per minute
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
liters per minute | 16.2 (4.5) | 14.9 (4.4) | 12.9 (4.6) | 20.6 (5.3)

7. Secondary Outcome: Change Between Week 44 and Week 0 Peak Expiratory Flow Rate (PEFR) Variability
Description: PEFR variability represents the relative change between the evening and morning PEFR measurements, so it could be a positive or negative number. It was measured daily during the 44-week treatment period. Specifically, the PEFR variability on a specific day is defined as 100% x (evening PEFR - morning PEFR)/{0.5*(evening PEFR + morning PEFR)}
Time Frame: PEFR variability was measured daily during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: relative change (AM and PM peak flow)
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
relative change (AM and PM peak flow) | 0.836 (0.51) | -0.043 (0.56) | 0.098 (0.53) | 0.894 (0.58)

8. Secondary Outcome: Change Between Week 44 and Week 0 in the Exhaled Nitric Oxide (eNO) Measured in Parts Per Billion
Time Frame: eNO was measured on seven occasions during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | Daily ICS + Rescue ICS | Daily ICS | Rescue ICS | Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
parts per billion | -0.08 (0.13) | 0.07 (0.11) | 0.58 (0.13) | 0.34 (0.14)

9. Secondary Outcome: Change Between Week 44 and Week 0 in the Asthma-specific Quality of Life Assessment
Description: The asthma-specific quality of life scale ranged from 1 (worst) to 7 (best)
Time Frame: The asthma-specific quality of life assessment was measured on seven occasions during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
units on a scale | 0.15 (0.09) | 0.07 (0.11) | 0.05 (0.15) | -0.03 (0.12)

10. Secondary Outcome: Change Between Week 44 and Week 0 in the Asthma Control Test (ACT)
Description: The ACT consisted of five questions, each ranging from 1 (worst) to 5 (best). The five questions were summed to yield an overall score that ranged from 5 (worst) to 25 (best).
Time Frame: The ACT was measured on seven occasions during the 44-week treatment period. The primary analysis constructed the change between week 44 and week 0.
Population: All randomized participants were included in the linear mixed-effects model analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Number analyzed (Participants) | 71 | 72 | 71 | 74
units on a scale | 0.17 (0.47) | -0.15 (0.46) | -0.57 (0.49) | -0.76 (54)

ADVERSE EVENTS:
Time Frame: 1 year
Description: does not differ from the clinicaltrials.gov definitions
Arm/Group | A: Daily ICS + Rescue ICS | B: Daily ICS | C: Rescue ICS | D: Placebo
Serious Adverse Events (participants affected / at risk) | 4/71 | 2/72 | 6/71 | 17/74
Other Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/71 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Daily ICS + Rescue ICS (N=71) | B: Daily ICS (N=72) | C: Rescue ICS (N=71) | D: Placebo (N=74)
Treatment Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 6 (6) | 17 (17) — Treatment failure was defined as the requirement for a second dose of prednisone within any 6-month period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No